CLINICAL TRIAL: NCT02189876
Title: Reducing HIV/STD Risk in African American Women With At-Risk Male Partners
Brief Title: Females of African American Legacy Empowering Self (FemAALES)
Acronym: FemAALES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of California, Los Angeles (Other); St. John's Well Child & Family Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MD-13-010; P20MD000182 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-07-15 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: HIV
Keywords: HIV Prevention; Behavioral Intervention; Condom Use; African American; Sexually Transmitted Disease; Sexually Transmitted Infection; Internet
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FemAALES (Experimental): Females of African American Legacy Empowering Self Intervention. A nine session, theoretically grounded small group intervention.
  Interventions: Behavioral: Standard of Care; Behavioral: FemAALES
- Standard of Care (Active Comparator): A one-time STD/family planning testing and counseling session provided to all study participants.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Standard of Care — All participants will be provided a STD/HIV pre-test counseling session. This session will be provided by either certified project staff or clinical staff at a Los Angeles clinic that conduct State of CA Fam Pact services for patients who are of child bearing age, including our current study partner St. John's Well Child and Family Center and our former study partner, JWCH (John Wesley Community Health) Institute-Wesley Health Center Clinics. Following the counseling session, the participant will be asked to provide a sample of urine to test for Chlamydia and Gonorrhea.
Behavioral: FemAALES — Women will attend 9 small group sessions over 4 weeks. Three of these sessions will focus specifically on participants learning to use a computer, set up an email account, communicate with the team and the group using the Internet, and developing a prevention message for display on project website and social media accounts. The other 6 sessions will include discussions on the following topics: being a Black woman in American, Black history, assessing personal health, changing current behaviors, HIV/AIDS information, and education, self-empowerment, communication skills, reasons to change, and goal setting.
  Arms: FemAALES

SUMMARY:
The FemAALES Project is a community collaborative two-arm intervention designed to prevent HIV (human immunodeficiency) and STD (sexually transmitted disease) infection and transmission among African American women and men by reducing sexual risk factors and enhancing sexual negotiation skills. The team of investigators is a collaboration of researchers and community service providers who are committed to developing prevention interventions that employ holistic and culturally relevant approaches. This includes recognizing the impact of forces such as racism, sexism, and gender expectations on individual behavior and relationship dynamics in African American communities. Specifically, the investigators hypothesis is that compared to the control condition the FemAALES intervention arm will reduce risky sexual behavior and STI (sexually transmitted infection) incidence and will increase condom self-efficacy and risk behavior communication with sexual partners.

DETAILED DESCRIPTION:
Two thirds of female HIV/AIDS cases occur in Black women and an estimated 76% of these are attributed to heterosexual contact. HIV is the third-leading killer of Black women ages 25-44, and STI associated morbidity may contribute to racial disparities in cervical cancer, adverse pregnancy outcomes, and infant mortality.

The investigators propose to test the efficacy of the FemAALES of African American Legacy Empowering Self Intervention in a population of adult Black/African American women who have either no health insurance or a public/subsidized form of health insurance against a Control or "Standard of Care" arm involving family planning and STI counseling.

In addition, the investigators will explore the impact of the FemAALES intervention on the use of new media for social support and networking, obtaining health information, and identifying resources and services. FemAALES incorporates cultural contextual, and partnership issues and promotes access to resources not readily available to this population. FemAALES curriculum is guided by the Theory of Reasoned Action and Planning and Critical Thinking and Cultural Affirmation Model developed by a collaborating community-based organization.

The primary specific aims are to:

1. Determine the impact of the FemAALES of African American Legacy Empowering Self (FemAALES II) on HIV risk factors including:

   1. number of sex partners
   2. unprotected anal/vaginal sex
   3. incidence of bacterial STIs
2. Determine the impact of the FemAALES interventions on psychosocial outcomes, including self-efficacy for safer sex negotiation and discussions with partners regarding HIV/STI testing and risk

   * Hypothesis 1: Compared to the control, FemAALES will reduce the number of vaginal/anal sex partners and number of episodes of unprotected intercourse at 3months and 9 months post intervention
   * Hypothesis 2: Compared to the control, FemAALES will reduce the incidence of gonorrhea and chlamydia
   * Hypothesis 3: Compared to the control, FemAALES will improve self-efficacy for condom negotiation
   * Hypothesis 4: Compared to the control. FemAALES will increase the proportion of women who have discussions regarding sexual and drug use risk factors with their sexual partners.

A third, exploratory aim, is to assess the impact of the FemAALES intervention on the use of new social media for social support and networking, obtaining health information and identifying resources and services.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* self-identifies as Black/African American
* 18 years of age or older
* English speaking
* has had unprotected vaginal or anal sex in the last 90 days
* any male partner in the last 90 days has done one or more of the following: had sex with a man; had sex with a male-to-female transgender; used crack cocaine, heroin, or methamphetamines; been incarcerated for more than 6 months; had sex with other female partners during the relationship; OR - a male partner in the last 90 days has an unknown sexual history
* publicly funded or public subsidized health insurance

Exclusion Criteria:

* participated in a small group HIV prevention program in the past 12 months, participated in HARRP program in the past 12 months, has private insurance, refuses chlamydia or gonorrhea test at baseline,

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 256 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in number of sex partners from baseline | 3 and 9 months
  Determine the impact of the FemAALES intervention compared to the control condition on the number of vaginal and anal sex partners in the prior 90 days .
Change in frequency of unprotected sex from baseline. | 3 and 9 months
  Determine the impact of the FemAALES interventions compared to the control condition on the number of vaginal or anal sex acts reported without condoms in the prior 90 days.
Change in bacterial STDs from baseline | 9 months
  Examine the impact of the FemAALES interventions compared to the control condition on the incidence of gonorrhea and chlamydia.

SECONDARY OUTCOMES:
Change in Safer Sex Negotiation Skills and Behaviors | 3 and 9 months
  Determine the impact of the FemAALES conditions compared to the control condition on psychosocial outcomes, including self-efficacy for safer sex negotiation and discussions regarding HIV/STI risk with sexual partners.

OTHER OUTCOMES:
Intervention Effect on Use of New Media | 9 months
  Determine the impact of the FemAALES intervention on the frequency and types of use of new media for social support, health information, and identifying resources.

CONTACTS AND LOCATIONS:
Overall Officials: Nina T Harawa, Ph.D, MPH, Principal Investigator — Charles Drew University; Martin Shapiro, MD Ph.D MPH, Principal Investigator — University of California, Los Angeles; Samuel Gonzalez, MS, Principal Investigator — St. John's Well Child and Family Center
Locations (2):
- United States (2):
  - St. John's Well Child and Family Center, Los Angeles, California
  - Charles Drew University of Medicine and Science, Los Angeles, California

REFERENCES:
- [Derived] Adeyeba MO, Montazeri Q, Bivens-Davis T, Schrode KM, Harawa NT. Reducing Human Immunodeficiency Virus and Sexually Transmitted Infections Risk in African American Women with At-Risk Male Partners: A Randomized Trial. J Womens Health (Larchmt). 2023 Mar;32(3):311-322. doi: 10.1089/jwh.2022.0194. Epub 2022 Dec 14. PMID 36520613